CLINICAL TRIAL: NCT00418470
Title: Prolonging the Duration on Site of Short Peripheral Venous Catheters Used to Administer Intravenous Antibiotics in Cystic Fibrosis Adults. Randomized Controlled Trial on the Effect of Different Concentrations of Antibiotic in Normal Saline
Brief Title: Prolonging the Duration of Peripheral Venous Catheters in Cystic Fibrosis People
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: impossibility to find volunteers
Sponsor: University of Florence (Other)
Collaborators: Italian Cystic Fibrosis Research Foundation (Other); Ospedale Meyer (Other)
Responsible Party: Principal Investigator, Filippo Festini, Associate Professor, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FFC #19/2006
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis; Phlebitis
Keywords: Cystic fibrosis; Catheterization, peripheral; Phlebitis; Anti-Bacterial Agents; Osmolar Concentration
MeSH Terms: conditions — Cystic Fibrosis; Phlebitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Higher concentration of antibiotic in NS
  Interventions: Procedure: regular dilution of antibiotic in NS
- B (Experimental): Lower concentration of antibiotic in NS
  Interventions: Procedure: higher dilution of antibiotic in NS

INTERVENTIONS:
Procedure: regular dilution of antibiotic in NS — IV administration of ceftazidime tid diluted in regular NS volume
  Arms: A
Procedure: higher dilution of antibiotic in NS — IV administration of ceftazidime tid diluted in larger NS volume
  Arms: B

SUMMARY:
Patients with cystic fibrosis (CF) need to frequently undergo courses of IV antibiotic therapy. To avoid a high number of venipunctures peripheral venous catheters (SPVC) or cannulas are used. Because of the irritant action of the drugs used, SPVC's often do not last for the whole antibiotic course (usually of two weeks) and the patient has to be punctured again for the insertion of a new IV line. With the passing of time the veins are more difficult to be found. An alternative to the use of a cannulas is the surgical insertion of a central venous catheter. This intervention may have contraindications or, specially in adolescents, cause unacceptable alterations of the body image.

The aim of this study is to find a way to prolong the duration of the SPVC used by CF patients during antibiotic courses avoiding the irritation of the vein or a phlebitis.

Design of the study: randomized controlled trial. The study will see a collaboration of nurses, physicians and technicians of the Tuscan CF Centre.

The patients that will participate at the study will be randomly assigned to one of the two groups: one group will receive the antibiotics prescribed according to the maximal dilution suggested by the pharmaceutical company, the other will receive a much higher dilution (i.e. a higher volume of Normal Saline), but the time of administration will be the same.

The assessment will regard: the level of inflammation of the vein (with a special visual scale) and the duration of the SPVC.

The hypothesis that is to be proved is that diluting the antibiotic in a higher volume of Normal Saline it is possible to delay or prevent the irritation of the vein and the onset of a phlebitis.

In case that the hypothesis will be confirmed by this study an easy, secure, low cost and immediately available system will be available to reduce the number of venipunctures necessary to complete a course of IV antibiotics.

DETAILED DESCRIPTION:
Background

Cystic Fibrosis (CF) is a common genetic disease which affects, among other organs, the respiratory tree. The major cause of mortality and morbidity in CF are pulmonary infections caused by a limited number of bacteria, in particular gram negative bacteria such as Pseudomonas aeruginosa (PA) and Burkholderia cepacia complex (BCC) which cause frequent clinically acute pulmonary infections.

Current figures show that 57.3% of patient have their lungs infected by PA and 2.9% of them have their lungs infected by BCC (1). To fight pulmonary exacerbations, patients frequently have to undergo antibiotic treatments, which often cannot be given orally or by aerosol but have to be administered intravenously (IV). Some CF Centers have also adopted a treatment protocol for patients chronically infected by respiratory pathogens in which a prophylactic IV course of antibiotic is routinely given every 3 months even in the absence of clinical symptoms of pulmonary exacerbations (2) An IV course of antibiotic treatment should be continued for at least 10 days but usually it lasts 2 weeks (3). Completing it would therefore require doing numerous venipunctures to a patient. In the USA, during 2004 some 45% of patients aged 18 to 30 required at least 1 IV antibiotic course, about 25% 2 IKV course and 15% 3 courses or more (1). This IV treatment regime brings a relevant burden of pain, anxiety and a worsening of quality of life (4). In order to reduce the number of venipunctures needed for an antibiotic course, several intravenous indwelling devices have been used to administer antibiotic infusion.

Some of these venous catheters are inserted in a central vessel. Among them, port caths and Groshong or Broviac type Central catheters, Midline catheters are those most commonly used (5-9). They are intended to last from several weeks to years. Their insertion requires a surgical intervention. Such an invasive intervention may not be sometimes indicated due to the patient's clinical condition. Moreover, the presence of a permanent device may influence the patients' body image and autonomy, with negative consequences in the psychological condition of the patient, especially in adolescence (10). Also, systemic infections may occur (11), the permanent management of the device may result complicated (12-15) and it may influence the patient's day-to-day life. Recently, a high incidence of thrombosis related to the insertion of this kind of catheters has been described (16) The most commonly used type of IV device to administer antibiotics in CF is the short peripheral venous catheter (SPVC) or cannula (17, 18) which has been considered for long now the simplest, most easy-to-use and economic way for administering IV therapy in CF. The use of this device allows patients not to be punctured at every administration and to eventually perform the antibiotic course at home avoiding hospitalisation and therefore maintaining a relatively normal daily life. Moreover, compared to the previously described permanent devices, this one is less invasive, it does not require a surgical intervention to be inserted, and it is intended to be maintained only for the duration of the treatment.

In order to facilitate CF people's autonomy and to reduce the conditioning of their quality of life, The home administration of IV antibiotic has become increasingly common (17-21). In 2004, 20.1% of US CF patients received home IV treatment (1). Patients themselves and their relatives are often trained by CF Centers' Nurses on how to manage the administration of the antibiotic treatment on their own.

Typical responsibilities of the CF Center's Nursing Staff is to position the SPVC, to manage the venous access and the drug infusions, to evaluate the site of the cannula insertion and the drug administration, and to educate patients on possible complications (21-23).

During the course, patency of the venous access between one antibiotic administration and the following is achieved by flushing the catheter at the end of each infusion either with normal saline or with heparin solution.

With the passing of time, SPVC insertion might become increasingly difficult due to the repeated venous trauma, which may lead to the formation of thrombi and the progressive occlusion of the vein; (17).

Due to the particular respiratory pathogens (PA, BCC) affecting CF patients' lungs the doses of antibiotics are much higher than those administered to non-CF patients with pneumonia. Even though it sensibly lowers the risk of infectious problems, the IV administration of such high doses of antibiotics, may irritate the veins' tunica intima and cause a phlebitis which may occlude the vein and therefore interrupt the vein's patency. Indeed, it is well established that the infusion of antibiotics and other irritant substances frequently cause iatrogenic phlebitis (24-28). Other factors have been discussed as risk factors for the onset of phlebitis and to a short duration of the SPVC (29); among others, the movement of the patient, his/her age, the type of SPVC, the type of dressing used, the site of insertion (30) the blood count, (25).

The onset of phlebitis oblige healthcare providers to the repositioning of the venous catheter in another site and to cause to the patient further suffering, pain and anxiety. Although scarcely investigated, the problem of reducing the amount of venipunctures and pain in CF patients is clinically important. A recent study by our research group has examined the recalls of adult CF patients about the invasive procedures received in childhood (31). The study has evidenced that repeated venipunctures imply an additional worsening of their quality of life and may influence the CF child future compliance to treatments.

So far only a few studies have investigated an effective way to prolong the duration of SPVCs used without causing a phlebitis, but they are substantially inconclusive (32,33) On the basis of the existing studies, it can be hypothesised that the volume of fluid in which the antibiotic is diluted, and consequently its concentration, may affect the veins' tunica intima irritation.

Specific Aims and Rationale

This study aims at investigating whether a different concentration of the prescribed dose of antibiotic in the infusate during intravenous administrations influences the inflammation of the vessels and the consequent duration of SPVCs in patients with CF undergoing antibiotic courses.

For each antibiotic to be administered IV, the producer, besides the type of infusate, provides also a suggested maximum concentration or a concentration range.

Theoretically it is possible to reduce the vessel's irritation by keeping the quantity of drug and the time of infusion constant, but diluting the prescribed amount of antibiotic in a larger volume of infusate, in a given interval of time. This would lead to a smaller number of drug molecules acting as irritants on the tunica intima.

Therefore, the aim of the study is to verify the hypothesis that a greater volume of infusate for constant amounts of drug dose and time, reduces the irritation of the vessel's tunica intima caused by the antibiotic and allows a longer patency of the vein and a longer use of the SPVC.

We will compare the outcomes of two different concentrations of antibiotic in Normal Saline, which is the mostly used infusate for IV administration of antibiotics. The type of the prescribed antibiotic and the time of infusion will stay the same. The CF center specialist physician will continue to prescribe drugs as usual, according to intern protocols and to patients' clinical conditions.

The eventual purpose of the study is to reduce patients' distress and discomfort when they are obliged to undergo antibiotic treatments which need invasive procedures. Indeed, if the tested hypothesis would be confirmed, simply increasing the volume of normal saline in which the antibiotic is diluted would lead to less vein irritation, lower incidence of phlebitis and a longer permanence of the SPVC used for an IV antibiotic course. This would imply a reduction of the number of venepunctures needed to complete an IV antibiotic course and a reduction of patient discomfort and pain.

Also, if the tested hypothesis would be confirmed, the solution proposed would be immediately applicable to the clinical practice, since it would not require any authorization process. Also, it would be of little expense and completely safe, unless any contraindications exists to the infusion of a higher volume of Normal Saline Besides this, CF Centers' Health Care Providers might have a simple, safe and relatively low-cost method to prolong the duration on site of a IV antibiotic course and to reduce the number of venepunctures given to the patient.

Preliminary results

Recently this same group of researchers has carried out an observational study, partially retrospective and partially prospective (34-36). We studied 87 SPVCs inserted to 36 patients in 56 IV antibiotic treatment cycles in a period of 6 months (mean duration 8.3 days). It has been evidenced that the gauge of the SPVC and the number of daily administrations are significantly correlated to the duration on site of the cannula. In particular, SPVCs with a larger gauge (G22) had longer mean duration than smaller (G24) SPVCs (9.6 days vs. 7.2 days, p=0.03) SPVCs used for antibiotic courses in which the antibiotic daily dose was divided into 3 administrations had a longer mean duration (10.3 days) than those used in courses in which the daily dose was divided into 2 administrations (6.5 days, p=0.001).

According to this study, other factors such as patients' age, the brand of the cannula, the health care professional who inserted the cannula, the site of insertion (dominating or non dominating arm), and the concurrent administration of oral anti-inflammatory drugs do not seem to influence the duration of the SPVC on site. The results of the study lead the researchers to hypothesise that the concentration of the antibiotic infusion i.e. its dilution might have an impact on the local inflammation of the vessel. Indeed, since each single administration was administered in the same infusion volume of 100 ml, the patients who had received the daily antibiotic dose divided in 3 administrations had received the same daily antibiotic dose diluted in a higher volume of fluids both daily and at each administration.

The study group is composed by Nurses, Physician and a Technician with a long experience in CF research. The group has carried out also other studies aimed at finding ways o that cures received by patients have as least impact as possible on their quality of life. In particular the study group's interest has focused on the issue of pain in CF patients (31, 37, 38).

Experimental Plan

Study design: Randomized controlled non-blinded clinical trial. The study will confront the effect of two different antibiotic concentrations administered IV on the inflammation of vein and on the duration in situ of the inserted SPVC.

The assignment of patients to one group or the other will be done by randomization. Randomization will be launched by a researcher blind in regards to patients. Data analysis will be done by a researcher blind in regards to patients.

The study will not influence the usual course of therapeutic treatment chosen by the specialized physician of the CF center. The only experimental variable will be the concentration of the dose of antibiotic prescribed by the physician in the infusate, or the volume of fluids needed to infuse the antibiotic.

In the aim of reducing the number of possible confounding variables, age range of the patients, SPVC gauge and brand, type of dressing, scales used for the evaluation of irritation and infiltration, type of antibiotics used, time of infusion, number of attempts for SPVC insertion will be standardized.

Authorization by the Ethic Committee of the Meyer Children Hospital has been obtained.

Subjects included to the study will sign an informed consent and the consent to treat their personal data. They will receive written information on the study.

Data will be analyzed and presented in aggregated form and by no means it will be possible to retrace the subjects to whom the data refer.

Subjects, Materials and Methods

This is a multidisciplinary study with participation of Nurse researchers, and Physician researchers They will participate in the study according to their own field of professional competences and legal responsibilities as described in the laws in force in Italy. In particular, Physicians will make diagnoses and order prescriptions and nurses will administer therapy, choose and use the most appropriate IV devices according to the clinical condition of the patient, notice and assess sign and symptoms with the use of validated scales, educate and instruct the patients on the therapy. Patients recruitment to the study will be done by the Physician and the Nurse together by assessing the fulfilment of inclusion criteria and by informing the patient.

The Nurses participating in the study will all be in possess of the qualification to practise the profession and of the graduate degree in Nursing or equivalent and will be instructed by the principal investigator in regards to the use of the assessment scales used in the study, the participants' inclusion criteria and the research protocol.

Inclusion criteria

To be included in the study subjects need to fulfil the following requirements:

* diagnosis of cystic fibrosis, made accordingly to the Cystic Fibrosis Foundation Guideline (Rosenstein BJ. J Pediatr 1998;132: 589-595)
* age of 18 years or more and ability to consciously express owns informed consent.
* have a prescription done by one of the CF Centre specialist Physicians of an IV antibiotic course of the foreseen duration of 2 weeks, due to a pulmonary exacerbation, with the association of ceftazidime 3 times daily and tobramycin once daily diluted in Normal Saline.
* absence of clinical conditions that contraindicate the administration of 350ml of Normal Saline in 30 minutes 3 times daily and of 400ml of Normal Saline in 40 minutes.
* no simultaneous anti-inflammatory therapy administered orally, IM or IV
* 30 days have passed from the end of the previous course.
* the IV course will be given to the subject as an inpatient, and he or she will be admitted to our hospital

The two experimental groups will have the following treatment:

Group A: Ceftazidime will be infused diluted in Normal Saline at the maximum suggested concentration of 40mg per ml of infusate. Time of infusion: 30 minutes.

Group B: Ceftazidime will be infused diluted in Normal Saline at the concentration of 10mg per ml of infusate. Time of infusion: 30 minutes.

For both group Tobramycin will be infused diluted in Normal Saline at the concentration of 1mg per ml of infusate (i.e., one half of the maximum suggested concentration of 1mg per ml of infusate). Time of infusion: 40 minutes.

Measured outcomes will be:

* the irritation level of the first vein that is cannulated for the course. The assessment will be done utilizing the "Phlebitis Scale" of the Standard of Practice of the Intravenous Nurses Society (39). The Scale is described in the "Clinical Protocol" Section..
* the number of days that the first SPVC used for the treatment course stays in situ before removal.

For each of the two groups calculation will be done on:

The proportion of subjects who will score 0 or 1 on the "Phlebitis Scale" for each single day of observation (1st day, 2nd day… up to the 14th) The mean duration of the first SPVC inserted for the treatment course

Statistical Analysis

Differences between proportions will be analysed with the Chi-square test. Differences between means of in situ durations of SPVCs will be analysed using the Student t-test.

Statistical significance level is established at 95%.

The removal of the first SPVC inserted for the antibiotic course concludes the participation of the subject to the study. The SPVC will be removed in the following cases:

* At the end of the IV course
* If the phlebitis level is 2 or more on the "Phlebitis Scale"
* If the infiltration level is 1 or more on the "Infiltration Scale" of the Standard of Practice of the Intravenous Nurses Society (39). The Scale is described in the "Clinical Protocol" Section.
* If pain is rated 3 or more on a numeric pain scale from 0 to 10 (40). If the subject needs to prolong the antibiotic therapy for more than 14 days the participation of the subject to the study will be over after the 14th day.

The same subject can be readmitted to the study if 30 days have passed from the end of the previous course.

The subject is a drop-out if

* He or she asks to remove the SPVC or takes it away autonomously or decides to refuse therapy.
* The patient starts having contraindications to the volume of Normal Saline infused
* The patient starts taking anti-inflammatory drugs orally or IM or IV.
* Patient refuses the prescribed therapy for more than 3 administrations or for 2 consecutive administrations.
* One or both prescribed antibiotics are modified by the specialized physician of the CF Centre because of changed clinical conditions of the subject; modification of the dose of ceftazidime or tobramycin does not interrupt the participation to the study if the concentration of the infusate remains the same. If this is the case the volume of Normal Saline will be changed according to the new dose subscribed.
* The SPVC is used for taking a blood sample or for the injection of any drug other than ceftazidime and tobramycin.
* The prescribed concentration is not respected, even if this happens only one time.

The data on the level of inflammation of the vein taken up to the moment of drop out will be included in the analysis according to the intention to treat. The duration of the SPVC will not be taken into account.

Determining the sample numerosity

The CF Center of Tuscany takes care of 191 patients. 78 patients (41%) are adults and potentially recruitable for the study. All patients of the Tuscan Regional CF Center are seen in the Outpatients clinic regularly to evaluate clinical status and microbiology of respiratory tract secretions. According to the data found with the preliminary study done by this same group of research (34), the antibiotic courses that match the inclusion criteria for this study in one year will be about 50 in the Tuscan CF Centre of Florence.

To determine the numerosity of the sample for the t-test on the differences between means of SPVC durations, we fixed a power of the trial of 0.8. In the absence of reference measures, we hypothesise a minimum expected difference between the SPVC duration in the two experimental groups equal to that found in the preliminary study carried out by this research group (34) between patients who were given IV antibiotics 2 times a day and those who received them 3 times a day, that is, 3.8 days. Also, we hypothesize a standard deviation within each group equal to that found in the two groups of the preliminary study, that is, 5. On the basis of these expected values, the numerosity of the two experimental groups was determined in 30 for each group. Such number will be increased of a number of subjects equal to the number of drop-outs.

Randomization

A simple randomization method will be utilized. One of the participants of the research group will do the randomization and will have no other role in the study. He will be blind concerning patients and will not know neither their identity nor their clinical status. Every time that a patient will be recruited into the study by the researchers, the Physician and the Nurse that have done the recruitment will contact the researcher responsible for the randomization to communicate that a new patient has been included without giving any information on the patient. The person responsible for randomization will flip a 50 cent Euro coin into the air and will communicate the result. The recto of the coin (the one indicating the coin value) means inclusion into the Group A. The verso of the coin (the one with the national insign) means inclusion into the Group B. The person responsible for randomization will be reachable by telephone on a dedicated mobile phone during all the CF Center opening time.

The study will end when both groups will have reached the numerosity established a priori, plus the number of drop-outs.

Sequence or Timetable of the Project

January 2007: education of the Nurses and of the Physicians that work at the clinical aspects of the study (recruitment, cannulation, knowing of the research protocol and preparation of the expected concentrations; assessment of cannulation site and use of the scales, education of the patient); February 2007: beginning of the recruitment of patients and start of the study June 2007: first check of the recruited patients and of the quality of collected data October 2007: second check of recruited patients and of the quality of collected data Retraining of all persons who collaborate at the study by the Principal investigator.

February 2008: third check of the recruited patients and of the quality of collected data June 2008: fourth check of recruited patients and of the quality of collected data Retraining of all persons who collaborate at the study by the Principal investigator.

October 2008: fifth check of recruited patients and of the quality of collected data February 2009: 6th check of the recruited patients and of the quality of collected data Retraining of all persons who collaborate at the study by the Principal investigator.

June 2009: 7th check of recruited patients and of the quality of collected data November 2009: end of data collection. Insertion of paper data into a Microsoft Access 2000 database.

December 2009. Statistical analysis. Writing of final report. Paper sent for evaluation to a peer-reviewed scientific journal

Clinical protocols

Recruitment of patients In occasion of a patient's visit to the CF Center Outpatient Clinic, the Physician decides, on the basis of the clinical conditions of patient, of laboratory tests, of results of sputum culture and other instrumental and imaging diagnostic tests, whether he or she needs an antibiotic treatment, of what type and by which way of administration.

If the physician decides to prescribe an antibiotic, the inclusion criteria are verified. If all the criteria are satisfied, the subject is eligible for the inclusion in the study.

The patient will be invited to participate to the study and will be given the necessary information. After answering to all his/her questions, if the patient accepts the inclusion, the Physician and the Nurse will collect his/her written informed consent.

Subsequently the Nurse will call the researcher in charge of randomisation and will ask him the group to which the patient is assigned.

Subsequently, the Nurse will collect the initial data of the patient in the recruitment form. Then he will insert the SPVC.

Way of administration of treatment To administer the treatment only Gauge 22 SPVCs Intima BD will be used. Before the insertion of SPVC the use of a local anaesthetic cream will be proposed to the patient, if not clinically contraindicated.

Before insertion, the insertion site will be disinfected with Amukine 5% solution. Skin hair will not be removed.

After the insertion the SPVC will be fixed to the skin with a sterile transparent dressing.

The dressing will not be changed or taken away during the experimentation in order to avoid displacement of the cannula. The SPVC will be closed with a needleless lock cap for all assessed subjects.

Each infusion will be administered during a total of 70 minutes: 30 minutes for the ceftazidime and 40 minutes for the tobramycin. There will be no flushing between the first and the second antibiotic. At the end of each infusion, the cannula will be flushed with 1.5 ml of a heparin solution (25 U/ml in Normal Saline). During the experimentation the SPVC cannot be used for any other therapy nor for the taking of blood samples.

Preparation of the concentrations as for the research protocol:

Table 1 indicates the dilutions to be prepared for each single administration of ceftazidime, according to the prescribed dose Group A

* 2000 mg.... 50 ml
* 2500 mg.... 62,5 ml
* 3000 mg.... 75 ml

Group B

* 2000 mg.... 200 ml
* 2500 mg.... 250 ml
* 3000 mg.... 300 ml

Table 2 shows the dilution to prepare for every single administration of tobramycin, according to the prescribed dose.

Both groups

* 150 mg.... 75 ml
* 200 mg.... 100 ml
* 250 mg.... 125 ml
* 300 mg.... 150 ml
* 350 mg.... 175 ml
* 400 mg.... 200 ml

In order to facilitate the preparation of the antibiotics to infuse according to the concentrations shown by the research protocol, a pharmaceutical company will prepare Normal Saline bottles prefilled with the volumes needed for the study.

Clinical assessment

At the moment of recruitment in the study the following data will be collected:

Age and sex, FEV1 (percentage of the predicted), body mass index, PCR, microorganism in the sputum culture, number of attempts needed to insert the SPVC.

Every day, before the IV midday administration a researcher will assess:

1. The state of irritation of the vein in which the SPVC is inserted, using the "Phlebitis scale" of the Standard of Practice of the Intravenous Nurses Society (39), as follows Grade Clinical Criteria

   * Grade 0.... No symptoms
   * Grade 1.... Erythema at access site with or without pain
   * Grade 2.... Pain at access site with erythema and/or edema
   * Grade 3.... Pain at access site with erythema and/or edema. Streak formation. Palpable venous cord
   * Grade 4.... Pain at access site with erythema and/or edema. Streak formation. Palpable venous cord >1 inch in length. Purulent drainage
2. The state of infiltration of the vein in which the SPVC is inserted, using the "Infiltration scale" of the Standard of Practice of the Intravenous Nurses Society (39) As follows.

   * Grade 0.... No symptoms
   * Grade 1.... Skin blanched, edema <1 inch in any direction, cool to touch, with or without pain
   * Grade 2.... Skin blanched, edema 1-6 inches in any direction; cool to touch; with or without pain.
   * Grade 3.... Skin blanched, translucent; gross edema >6 inch in any direction; cool to touch; mild-moderate pain; possible numbness.
   * Grade 4.... Skin blanched, translucent; skin tight, leaking, skin discoloured, bruised, swollen; gross edema >6 inch in any direction; deep pitting tissue edema; circulatory impairment; moderate-severe pain;infiltration of any amount of blood product, irritant, or vesicant
3. The pain experienced locally by the patient using the numeric pain scale.
4. Adverse events, the physical activity performed and any other event related to the antibiotic course which may have occurred in the previous 24 hours, as described by the patient.

The researcher will ascertain, with questions and other checks, that in the previous 24 hours the dilution provided in the research protocol has been respected and that no violations of the protocol have occurred.

In rare cases, patients who have started the course as inpatients may continue it at their home, as described before (23). In these cases patients will be given a high resolution mobile videophone. The researcher will phone to the patient, will interview him and will assess the insertion site using the videophone. The validity of this kind of distance evaluation has been recently showed by a study performed on leg ulcers (41).

If the assessor scores the insertion site 2 or more in the "Phlebitis Scale", or 1 or more in the "Infiltration scale", or the patient reports a local pain of 3 or more in the pain numeric rating scale, the SPVC is removed and the observation of the subject in the study ends.

Quality controls

Every 4 months the Principal Investigator will verify the number of recruited patients and of the quality of collected data, analysing all the daily assessment forms. In case of drop-outs the number of patients to be recruited will be increased by an equal number of subjects.

Every 8 months the Principal Investigator will retrain all the collaborators involved in the study in particular with regard to: recruiting, vein cannulation, knowledge of the research protocol, preparation of antibiotic dilutions, use of scales, training of patient.

Safety

For this research we will not use any method or drug which deviate from the normal clinical practice; we will apply usual operational procedures for prevention of Clinical Risk approved for the Hospital by the Local Committee for Patient Safety and Clinical Risk Management, as provided by the Tuscan Regional Government Decree n. 1387/2004). Also, the Principal Investigator is a member of such Committee.

Adverse events relating to the participation to the study will be constantly monitored. A member of the study group will be always reachable by phone by patients for any problem that may occur during the study.

Data management and statistical analysis

Data will be stored in a Microsoft Access 2000 database. Statistical analysis will be performed by an independent free-lance Statistician, not belonging to the Researchers' Institution.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis, made accordingly to the Cystic Fibrosis Foundation Guideline (Rosenstein BJ. J Pediatr 1998;132: 589-595)
* age of 18 years or more and ability to consciously express owns informed consent.
* have a prescription done by one of the CF Centre specialist Physicians of an IV antibiotic course of the expected duration of 2 weeks, due to a pulmonary exacerbation, with the association of ceftazidime 3 times daily and tobramycin once daily diluted in Normal Saline.
* absence of clinical conditions that contraindicate the administration of 350ml of Normal Saline in 30 minutes 3 times daily and of 400ml of Normal Saline in 40 minutes.
* no simultaneous anti-inflammatory therapy administered orally, IM or IV
* 30 days have passed from the end of the previous course.
* The IV course will be given to the subject as an inpatient, and he or she will be admitted to our hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The irritation level of the first vein that is cannulated for the course assessed each day. The assessment will be done utilizing the "Phlebitis Scale" of the Standard of Practice of the Intravenous Nurses Society (Journal of Intravenous Nursing 2000; | once a day
The number of days that the first short peripheral venous catheter used for the treatment course stays in situ before removal | once a day

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Festini, RN, BA, BSN, Principal Investigator — University of Florence, Department of Pediatrics
Locations (1):
- Meyer Pediatric Hospital (Ospedale Pediatrico Meyer), Florence, Italy

REFERENCES:
- [Background] Cystic Fibrosis Foundation. Patient Registry 2004 Annual Report. Bethesda, Maryland
- [Background] Breen L, Aswani N. Elective versus symptomatic intravenous antibiotic therapy for cystic fibrosis. Cochrane Database Syst Rev. 2001;(4):CD002767. doi: 10.1002/14651858.CD002767. PMID 11687159
- [Background] Littlewood J, Bevan A, Commet G, Govan J. Antibiotic treatment for cystic fibrosis. Cystic Fibrosis Trust 2002. Bromley, UK
- [Background] Esmond G, Butler M, McCormack AM. Comparison of hospital and home intravenous antibiotic therapy in adults with cystic fibrosis. J Clin Nurs. 2006 Jan;15(1):52-60. doi: 10.1111/j.1365-2702.2005.01236.x. PMID 16390524
- [Background] Munck A, Malbezin S, Bloch J, Gerardin M, Lebourgeois M, Derelle J, Bremont F, Sermet I, Munck MR, Navarro J. Follow-up of 452 totally implantable vascular devices in cystic fibrosis patients. Eur Respir J. 2004 Mar;23(3):430-4. doi: 10.1183/09031936.04.00052504. PMID 15065834
- [Background] Gronowitz E, Strandner K, Herlitz K et all. A national Swedish survey of totally implantable venous access devices (TIVAD) in patients with Cystic Fibrosis (CF). J Cyst Fibros 2003;2:S72
- [Background] Tolomeo C, Mackey W. Peripherally inserted central catheters (PICCs) in the CF population: one center's experience. Pediatr Nurs. 2003 Sep-Oct;29(5):355-9. PMID 14651306
- [Background] Millar-Jones L, Goodchild MC. Peripheral long lines in cystic fibrosis. J Clin Pharm Ther. 1997 Feb;22(1):45-6. doi: 10.1046/j.1365-2710.1997.94075940.x. PMID 9292402
- [Background] Williams J, Smith HL, Woods CG, Weller PH. Silastic catheters for antibiotics in cystic fibrosis. Arch Dis Child. 1988 Jun;63(6):658-9. doi: 10.1136/adc.63.6.658. PMID 3389899
- [Background] Campbell WB, Elworthy S, Peerlinck I, Vanslembroek K, Bangur R, Stableforth D, Sheldon CD. Sites of implantation for central venous access devices (ports): a study of the experiences and preferences of patients. Eur J Vasc Endovasc Surg. 2004 Dec;28(6):642-4. doi: 10.1016/j.ejvs.2004.08.002. PMID 15531201
- [Background] Proesmans M, Boulanger L, De Boeck K. Complications with indwelling catheters in CF patients followed at the universital hospital in Leuven (Belgium). J Cyst Fibros 2002;S172-S173.
- [Background] Miall LS, Das A, Brownlee KG, Conway SP. Peripherally inserted central catheters in children with cystic fibrosis. Eight cases of difficult removal. J Infus Nurs. 2001 Sep-Oct;24(5):297-300. doi: 10.1097/00129804-200109000-00003. PMID 11575044
- [Background] Deerojanawong J, Sawyer SM, Fink AM, Stokes KB, Robertson CF. Totally implantable venous access devices in children with cystic fibrosis: incidence and type of complications. Thorax. 1998 Apr;53(4):285-9. doi: 10.1136/thx.53.4.285. PMID 9741372
- [Background] Rodgers HC, Liddle K, Nixon SJ, Innes JA, Greening AP. Totally implantable venous access devices in cystic fibrosis: complications and patients' opinions. Eur Respir J. 1998 Jul;12(1):217-20. doi: 10.1183/09031936.98.12010217. PMID 9701441
- [Background] Jacobs WR, Zaroukian MH. Coughing and central venous catheter dislodgement. JPEN J Parenter Enteral Nutr. 1991 Jul-Aug;15(4):491-3. doi: 10.1177/0148607191015004491. PMID 1823540
- [Background] Barker M, Thoenes D, Dohmen H, Friedrichs F, Pfannenstiel C, Heimann G. Prevalence of thrombophilia and catheter-related thrombosis in cystic fibrosis. Pediatr Pulmonol. 2005 Feb;39(2):156-61. doi: 10.1002/ppul.20158. PMID 15633202
- [Background] Strandvik B, Hjelte L, Malmborg AS, Widen B. Home intravenous antibiotic treatment of patients with cystic fibrosis. Acta Paediatr. 1992 Apr;81(4):340-4. doi: 10.1111/j.1651-2227.1992.tb12239.x. PMID 1606396
- [Background] Giron RM, Martinez A, Maiz L, Salcedo A, Beltran B, Martinez MT, Antelo C, Barrio I, Prados C, Cabanillas J, Ancochea J. [Home intravenous antibiotic treatments in cystic fibrosis units of Madrid]. Med Clin (Barc). 2004 May 8;122(17):648-52. doi: 10.1016/s0025-7753(04)74341-9. Spanish. PMID 15153343
- [Background] Salcedo A, Giron RM, Beltran B, Martinez A, Maiz L, Suarez L; Fundacion Sira Carrasco. [Consensus conference: home intravenous antibiotic treatment for cystic fibrosis. The Sira Carrasco Foundation. 26 April 2002]. Arch Bronconeumol. 2003 Oct;39(10):469-75. doi: 10.1016/s0300-2896(03)75430-1. No abstract available. Spanish. PMID 14533997
- [Background] Riethmueller J, Busch A, Damm V, Ziebach R, Stern M. Home and hospital antibiotic treatment prove similarly effective in cystic fibrosis. Infection. 2002 Dec;30(6):387-91. doi: 10.1007/s15010-002-2095-0. PMID 12478330
- [Background] Kerem E, Conway S, Elborn S, Heijerman H; Consensus Committee. Standards of care for patients with cystic fibrosis: a European consensus. J Cyst Fibros. 2005 Mar;4(1):7-26. doi: 10.1016/j.jcf.2004.12.002. No abstract available. PMID 15752677
- [Background] The UK CF Nurse Specialist Group. National consensus standards for the nursing management of cystic fibrosis. London, UK7 Cystic Fibrosis Trust; 2001.
- [Background] Duncan-Skingle F, Bramwell E. Cystic Fibrosis Home care. In: Hodson ME, Geddes DM. Cystic Fibrosis. Arnold, London, 2000.
- [Background] Regueiro Pose MA, Souto Rodriguez B, Iglesias Marono M, Outon Fernandez I, Cambeiro Nunez J, Pertega Diaz S, Pita Fernandez S. [Peripheral venous catheters: incidence of phlebitis and its determining factors]. Rev Enferm. 2005 Oct;28(10):21-8. Spanish. PMID 16304830
- [Background] Monreal M, Quilez F, Rey-Joly C, Rodriguez S, Sopena N, Neira C, Roca J. Infusion phlebitis in patients with acute pneumonia: a prospective study. Chest. 1999 Jun;115(6):1576-80. doi: 10.1378/chest.115.6.1576. PMID 10378551
- [Background] Tager IB, Ginsberg MB, Ellis SE, Walsh NE, Dupont I, Simchen E, Faich GA. An epidemiologic study of the risks associated with peripheral intravenous catheters. Am J Epidemiol. 1983 Dec;118(6):839-51. doi: 10.1093/oxfordjournals.aje.a113702. PMID 6650485
- [Background] Falchuk KH, Peterson L, McNeil BJ. Microparticulate-induced phlebitis. Its prevention by in-line filtration. N Engl J Med. 1985 Jan 10;312(2):78-82. doi: 10.1056/NEJM198501103120203. PMID 3880597
- [Background] Hessov I, Allen J, Arendt K, Gravholt L. Infusion thrombophlebitis in a surgical department. Acta Chir Scand. 1977;143(3):151-4. PMID 411297
- [Background] Lanbeck P, Odenholt I, Paulsen O. Perception of risk factors for infusion phlebitis among Swedish nurses: a questionnaire study. J Infus Nurs. 2004 Jan-Feb;27(1):25-30. doi: 10.1097/00129804-200401000-00004. PMID 14734984
- [Background] Brandt CT. [Phlebitis due to venous catheters. Causes and occurrence]. Ugeskr Laeger. 2000 Aug 21;162(34):4531-4. Danish. PMID 10981220
- [Background] Neri S, Allegretti N, Vignoli N, FESTINI F. Perception of pain and fear related to invasive procedures in children with cystic fibrosis: a study using CF adults recalls. J Cyst Fibros 2006; 5 (suppl1): 91.
- [Background] Richards C, Millar-Jones L, Alfaham M. Assessment of in-line filters to prolong the life of intravenous cannulae in cystic fibrosis patients. J Clin Pharm Ther. 1995 Jun;20(3):165-6. doi: 10.1111/j.1365-2710.1995.tb00643.x. PMID 7593378
- [Background] Roberts GW, Holmes MD, Staugas RE, Day RA, Finlay CF, Pitcher A. Peripheral intravenous line survival and phlebitis prevention in patients receiving intravenous antibiotics: heparin/hydrocortisone versus in-line filters. Ann Pharmacother. 1994 Jan;28(1):11-6. doi: 10.1177/106002809402800101. PMID 8123947
- [Background] Festini F, Beneventi R, Vignoli N, Allegretti N, Rontini I, Campigatto E, Grondoni G, Sanasi S, Bongini G. [Factors that influence the duration of peripheral venous catheters used to antibiotic therapy in Cystic Fibrosis patients: results of a study]. Assist Inferm Ric. 2005 Apr-Jun;24(2):91-6. Italian. PMID 16218243
- [Background] FESTINI F, Beneventi R, Allegretti N, Vignoli N, Chiarelli F. Does oral anti.inflammatory therapy influence the duration of peripheral venous catheters used for IV antibiotic cycles in cystic fibrosis patients ? Pediatr Pulmonol 2005; Suppl 28: 359-360.
- [Background] Festini F, Ballarin S, Codamo T, Doro R, Loganes C. Prevalence of pain in adults with cystic fibrosis. J Cyst Fibros. 2004 Mar;3(1):51-7. doi: 10.1016/j.jcf.2003.12.001. PMID 15463887
- [Background] Ballarin S, Codamo T, Doro R, Loganes C, FESTINI F. Pain in Italian Cystic Fibrosis adult patients: preliminary results of a national nurse led study. J of Cystic Fibrosis 2001; 1: 362.
- [Background] Alexander M (editor) Infusion Nursing Standard of Practice of the Intravenous Nurses Society. Journal of Intravenous Nursing 2000; 23. 6S.
- [Background] Hockenberry MJ. Wong's clinical manual of pediatric nursing. Mosby 2004, St Louis, Missouri.
- [Background] Braun RP, Vecchietti JL, Thomas L, Prins C, French LE, Gewirtzman AJ, Saurat JH, Salomon D. Telemedical wound care using a new generation of mobile telephones: a feasibility study. Arch Dermatol. 2005 Feb;141(2):254-8. doi: 10.1001/archderm.141.2.254. PMID 15724023